CLINICAL TRIAL: NCT02547831
Title: Tailored Beta-catenin Mutational Approach in Extra-abdominal Sporadic Desmoids Tumor Patients
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: INT 13/12
Record Dates: First submitted 2015-01-28; First posted 2015-09-11 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2015-09

CONDITIONS: Desmoid-type Fibromatosis
MeSH Terms: conditions — Desmoid Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational approach: Patients will be placed on wait and see approach and then shifted to specific treatment in case of progression
  Interventions: Other: Observational approach

INTERVENTIONS:
Other: Observational approach — Patients will be placed under wait and see approach without any specific treatment
  Other Names: Wait and see approach

SUMMARY:
This is a prospective, multicenter observational study under the umbrella of the ISG (Italian Sarcoma Group) evaluating local progression-free survival at 3 years of patients affected by extra-abdominal primary fibromatosis managed with front-line conservative approach and treated only in case of demonstrated progressive disease.

All patients included will be placed on wait and see approach and then shifted to treatment in case of documented radiological progressive disease.

For patient primarily evaluated for suspected desmoid tumor, a core-needle biopsy (eventually under CT/ultrasound guide) will be obtained for histological diagnosis and mutational analysis of CTNNB1 exon 3 (gene encoding Beta-catenin). If incisional biopsy or surgical procedure has done elsewhere, samples will be requested for histological confirmation and mutational analysis (centralization at the investigators Institution).

In case of progression at 3 months, defined as tumor growth documented radiologically (by contrast enhanced MRI) by Response Evaluation Criteria in Solid Tumors (RECIST), administered treatments will be proposed and then registered in the clinical database.The choice of the treatment and eventually the possibility of continuation of " surveillance only" will be at the discretion of Institution's Multidisciplinary Sarcoma Committee or as part of clinical trials with the consent of patient.

DETAILED DESCRIPTION:
This is a prospective, multicenter observational study under the umbrella of the ISG (Italian Sarcoma Group) evaluating local progression-free survival at 3 years of patients affected by extra-abdominal primary fibromatosis managed with front-line conservative approach and treated only in case of demonstrated progressive disease.

All patients included will be placed on wait and see approach and then shifted to treatment in case of documented radiological progressive disease.

For patient primarily evaluated for suspected desmoid tumor, a core-needle biopsy (eventually under CT/ultrasound guide) will be obtained for histological diagnosis and mutational analysis of CTNNB1 exon 3 (gene encoding Beta-catenin). If incisional biopsy or surgical procedure has done elsewhere, samples will be requested for histological confirmation and mutational analysis (centralization at our Institution) and in selected cases a new biopsy will be obtained.

In case of progression at 3 months, defined as tumor growth documented radiologically (by contrast enhanced MRI) by Response Evaluation Criteria in Solid Tumors (RECIST), administered treatments will be proposed and then registered in the clinical database (radiological evaluation will be centralized at Istituto Rizzoli, Bologna- Dr. Vandel).

Therapy will include the following options:

* Surgery
* Radiotherapy
* Medical treatment including hormonal therapy (e.g., tamoxifen, toremifene), low-dose chemotherapy (e.g.,methotrexate and vinorelbine/vinblastine), NSAIDs (e.g., celecoxib), and target therapy (Glivec)
* Combination The choice of the treatment and eventually the possibility of continuation of " surveillance only" will be at the discretion of Institution's Multidisciplinary Sarcoma Committee or as part of clinical trials with the consent of patient.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic forms
* No age limit (pediatric patients can be included)
* Extra abdominal fibromatosis primary or with previous inadequate resection (R2) of the extremities, chest/abdominal wall and head/neck
* Histological diagnosis according to the WHO criteria done on biopsy or surgical specimen by our pathologist
* Diagnostic radiological exam performed (contrast enhanced MRI- T1 and T2 weighted)
* Signed informed consent form
* Adequate compliance of the patients to the plan of follow-up

Exclusion Criteria:

* Controindication to MRI
* Familial-type desmoid
* Recurrence
* Extraabdominal primary fibromatosis resected with R0/R1 margins
* Patients on treatment for desmoid tumor
* Other malignancies within past 5 years, with exception of carcinoma in situ of cervix and basocellular skin cancers treated with eradicating intent
* Serious psychiatric disease that precludes informed consent or limits compliance
* Medical disease requesting treatment corresponding to one of the drugs currently use in desmoid tumor [hormonal therapy (e.g., tamoxifen/toremifene, low-dose chemotherapy (e.g., methotrexate and vinorelbine/vinblastine), NSAIDs (e.g., celecoxib), and target therapy (Glivec)]
* Impossibility to ensure adequate follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by extra-abdominal primary fibromatosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gronchi, MD, Principal Investigator — Fondazione IRCCS Istituto Tumori Milano
Locations (2):
- Italy (2):
  - Fondazione del Piemonte per l' Oncologia - IRCCS, Candiolo, Torino
  - Fondazione IRCCS Istituto Tumori Milano, Milan

REFERENCES:
- [Derived] Colombo C, Fiore M, Grignani G, Tolomeo F, Merlini A, Palassini E, Collini P, Stacchiotti S, Casali PG, Perrone F, Mariani L, Gronchi A. A Prospective Observational Study of Active Surveillance in Primary Desmoid Fibromatosis. Clin Cancer Res. 2022 Sep 15;28(18):4027-4032. doi: 10.1158/1078-0432.CCR-21-4205. PMID 35247923